CLINICAL TRIAL: NCT06697769
Title: The Effect of Breastfeeding Experience Presented to Pregnant Women With Virtual Reality Glasses on Breastfeeding Self-efficacy and Breastfeeding Motivation: A Randomized Controlled Trial
Brief Title: The Effect of Breastfeeding Experience With Virtual Reality Glasses on Breastfeeding Self-efficacy and Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Nebahat ÖZERDOĞAN, Prof. Dr., Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Nebahat ÖZERDOĞAN
Record Dates: First submitted 2024-11-13; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Virtual Reality; Breastfeeding
Keywords: breastfeeding; virtual reality; pregnant women
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: A randomized study with a control and intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Individual standard breastfeeding education was provided. After the training, they experienced the first breastfeeding simulation in a hospital environment for 5 minutes with virtual reality glasses. A week later (37. during the gestational week), they experienced the second breastfeeding simulation in a home environment for 5 minutes with virtual reality glasses. They completed the Prenatal Breastfeeding Self-efficacy Scale (final test). Finally, 1 after giving birth. and 2. they completed the Primiparous Breastfeeding Motivation Scale between months. Opinions were obtained from pregnant women who wanted to express their opinions about the virtual reality glasses breastfeeding simulation experiences.
  Interventions: Other: virtual reality
- Control (No Intervention): Before starting the study, pregnant women who will be included in the control group according to the inclusion criteria and randomization were informed by the researcher about the study. At the beginning of the study, the control group (36. during the week of pregnancy) pregnant women filled out the Socio-Demographic and Pregnancy Information Form, Prenatal Breastfeeding Self-efficacy Scale (pre-test). Then, individual standard breastfeeding training was given. A week later (37. during the week of pregnancy), they completed the Prenatal Breastfeeding Self-efficacy Scale (final test). Finally, 1 after giving birth. and 2. they completed the Primiparous Breastfeeding Motivation Scale between months.

INTERVENTIONS:
Other: virtual reality — breastfeeding simulation with virtual reality glasses
  Arms: Virtual Reality

SUMMARY:
In this study, it was aimed to investigate the effect of breastfeeding experience on breastfeeding self-efficacy and motivation in women with virtual reality simulation. The main question it aims to answer is:

Is breastfeeding experience with virtual reality glasses effective in increasing breastfeeding self-efficacy and motivation? They completed the Socio-Demographic and Pregnancy Information Form and the Prenatal Breastfeeding Self-efficacy Scale. Standard breastfeeding training was given. The application group also experienced breastfeeding with a virtual reality simulation. At the end of the application, they filled out the Prenatal Breastfeeding Self-efficacy Scale again. They completed the postpartum Primiparous Breastfeeding Motivation Scale.

DETAILED DESCRIPTION:
Aim: In this study, it was aimed to investigate the effect of breastfeeding experience on breastfeeding self-efficacy and motivation in women with virtual reality simulation.

Desing: This study is a randomized controlled trial. Method: A total of 52 people were included in the study, 26 in the control group and 26 in the intervention group. They completed the Socio-Demographic and Pregnancy Information Form and the Prenatal Breastfeeding Self-efficacy Scale. Standard breastfeeding training was given. The application group also experienced breastfeeding with a virtual reality simulation. At the end of the application, they filled out the Prenatal Breastfeeding Self-efficacy Scale again. They completed the postpartum Primiparous Breastfeeding Motivation Scale.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 and over,
* Which is the primiparous,
* 36. during the week of pregnancy,
* Women whose pregnancy is not in the risky group,
* The person who knows how to read and write,
* Without visual and auditory disabilities,
* There is no breastfeeding barrier,
* Pregnant women who have experienced virtual reality breastfeeding experience and filled out the survey forms completely have been included in the research.

Exclusion Criteria:

* Individuals who did not meet the inclusion criteria were not included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Prenatal Breastfeeding Self-Efficacy Scale | The breastfeeding experience with virtual reality glasses lasted 5 minutes. The intervention was repeated a second time a week later over a 5-minute period. After two weeks of intervention, the last Breastfeeding Self-efficacy Scale test was applied.
  The Prenatal Breastfeeding Self-Efficacy Scale was developed by Wells and colleagues in 2006. The validity and reliability study of the scale in Turkish was conducted by Aydın and Pasinlioğlu in 2018. The scale consists of 20 items and is 5-point likert type. The lowest score to be taken from the scale is 20 and the highest score is 100. An increase in the score obtained from the scale indicates an increase in the perception of breastfeeding self-efficacy. The Cronbach Alpha value of the scale is 0.85.

SECONDARY OUTCOMES:
Primipar Breastfeeding Motivation Scale | The scale was completed up to two months after delivery.
  The adaptation of the Breastfeeding Motivation Scale developed by Kestler-Peleg (2015) to Turkish was carried out by Mızrak and Özerdogan in 2017. The scale for primiparous mothers consists of 23 items. Items are scored as 1, 2, 3, 4. The total score is not taken from the scale. As the score obtained from the sub-dimension of the scale increases, the motivation representing that sub-dimension also increases. The Cronbach alpha value of the scale is 0.887.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru ERTAŞ, Study Chair — ebru.ertas@ksbu.edu.tr; Feride ÇEVİK, Study Chair — feride.cevik@ksbu.edu.tr
Locations (1):
- Eskisehir Orhangazi Family Health Center, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang K, Gerling K, Chen W, Geurts L. Information and Communication Systems to Tackle Barriers to Breastfeeding: Systematic Search and Review. J Med Internet Res. 2019 Sep 27;21(9):e13947. doi: 10.2196/13947. PMID 31573903